CLINICAL TRIAL: NCT07203703
Title: Accuracy of Diagnostic Mounting With Jaw Tracking Device Versus Conventional Mounting Technique on Occlusal Contact Points in Dentate Patients: A Diagnostic Test Accuracy Study
Brief Title: Comparing Jaw Tracking and Traditional Methods for Measuring Bite Accuracy in Patients With Teeth
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Omer Abdelmagid (Other)
Responsible Party: Sponsor-Investigator, Omer Abdelmagid, Principal investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14422022455531
Record Dates: First submitted 2025-09-25; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Jaw Tracking
Keywords: Diagnostic Mounting; Jaw Tracking Device; Conventional Mounting Technique; Occlusal Contact Points

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Conventional Mounting Technique (Experimental)
  Interventions: Device: Jaw Tracking Device

INTERVENTIONS:
Device: Jaw Tracking Device — A jaw tracking device is a digital tool that records real-time jaw movements to accurately analyze occlusion and assist in virtual model mounting.

SUMMARY:
This study compares two methods used to measure how teeth come together (occlusal contacts) in patients who have natural teeth (dentate patients). The first method uses a modern jaw tracking device, while the second relies on the conventional mounting technique. The goal is to determine which method is more accurate for diagnosing bite alignment and contact points. This is a diagnostic test accuracy study, meaning it focuses on evaluating how well each technique performs in identifying the correct occlusal contacts.

DETAILED DESCRIPTION:
This study is a diagnostic test accuracy investigation aimed at comparing the precision of two different methods for diagnostic mounting in evaluating occlusal contact points in dentate patients (patients with natural teeth).

The two mounting techniques being compared are:

Jaw Tracking Device-Based Mounting This is a digital approach that utilizes a jaw tracking system to record the patient's mandibular movements accurately. The device captures dynamic jaw positions in real time, allowing for precise simulation of the patient's occlusion on an articulator or in a digital environment.

Conventional Mounting Technique This is the traditional, manual method using mechanical articulators. It typically involves facebow transfer and static bite records to mount the maxillary and mandibular casts in the assumed position. While widely used, this method may be prone to human error and variability.

The primary objective of the study is to assess and compare the accuracy of these two mounting techniques by examining how closely each one replicates the actual occlusal contact points observed intraorally. Occlusal contacts are critical in diagnosing and planning treatments in prosthodontics, orthodontics, and restorative dentistry.

By evaluating these contacts using both methods, the study aims to determine:

Which technique provides a more accurate representation of the patient's true occlusion.

The potential clinical implications of using a jaw tracking device over conventional methods.

Whether digital methods can improve diagnostic reliability and treatment outcomes in daily dental practice.

This study is expected to contribute to the growing body of evidence supporting digital technologies in dentistry, offering insights into their clinical accuracy and potential to replace or supplement traditional techniques.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 to 60 years Presence of full natural dentition (excluding third molars) No history of occlusal rehabilitation or major prosthodontic treatment

Exclusion Criteria:

Patients with missing teeth (excluding third molars) Patients with bruxism or other parafunctional habits History of orthodontic treatment in the past 2 years Inability to cooperate with diagnostic procedures patient below 18 years old

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of occlusal contact point detection as measured by comparing the contact points obtained from each mounting technique (jaw tracking device vs. conventional mounting) with the clinical intraoral occlusal contacts observed using articulating paper | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Nouran A Abdel Nabi, Professor, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: Yes
study protocol and statistical analysis
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 3 months
Access Criteria: will be with other investigator including who will work with systematic review, will provide the clinical study report with the documents above

REFERENCES:
- [Background] Tejo SK, Kumar AG, Kattimani VS, Desai PD, Nalla S, Chaitanya K K. A comparative evaluation of dimensional stability of three types of interocclusal recording materials-an in-vitro multi-centre study. Head Face Med. 2012 Oct 5;8:27. doi: 10.1186/1746-160X-8-27. PMID 23039395
- [Background] Rohrle O, Waddell JN, Foster KD, Saini H, Pullan AJ. Using a motion-capture system to record dynamic articulation for application in CAD/CAM software. J Prosthodont. 2009 Dec;18(8):703-10. doi: 10.1111/j.1532-849X.2009.00510.x. Epub 2009 Sep 14. PMID 19754645
- [Background] Pieper R. Digital impressions--easier than ever. Int J Comput Dent. 2009;12(1):47-52. English, German. PMID 19213360
- [Background] Kurbad A. Impression-free production techniques. Int J Comput Dent. 2011;14(1):59-66. English, German. PMID 21657126
- [Background] Kordass B. Clinical dental CAD/CAM--qualification for tomorrow's networked dentistry. Int J Comput Dent. 2010;13(1):3-6. No abstract available. English, German. PMID 20481287
- [Background] de Carvalho Ode T. A new fully adjustable articulator system and procedure. J Prosthet Dent. 1998 Sep;80(3):376-86. doi: 10.1016/s0022-3913(98)70141-6. PMID 9760374